CLINICAL TRIAL: NCT07051044
Title: Rapid Absorbance-based Detection of Inner Cheek Cell Abnormalities Using Light Spectroscopy for Risk Evaluation of Lung Cancer to Enable Critical Decision Support in Targeted Patient Populations
Acronym: RADICAL-REACT
Status: Recruiting | Type: Observational
Sponsor: Sierra Medical Ltd. (Industry)
Collaborators: Queen Alexandra Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: RADICAL-REACT
Record Dates: First submitted 2024-06-19; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cheek Swab taken from participants and processed onto an FTIR window and lab slides. Samples may be used for future testing or future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: AIR-DS — AIR-DS is a supportive, non-diagnostic, risk-indicating software that assists healthcare providers in the early detection and risk assessment of lung cancer in high-risk populations, aiming to improve the cost-effectiveness and accessibility of lung cancer screening. It is imperative to note that the efficacy of the AIR-DS may be affected by the completeness and accuracy of the input data. Hence, any missing data fields should be identified, as they could impact the risk assessment's accuracy.

SUMMARY:
Overview Sierra Medical is at the forefront of early detection of lung cancer by creating AIR-DS, a non-invasive early detection test. This innovative approach aims to significantly enhance the early identification of lung cancer, potentially catching it at its most treatable stages through a simple cheek swab.

How it works The effectiveness of AIR-DS stems from its ability to identify small biochemical changes in cells from the inner cheek. These biochemical changes can serve as early indicators of lung cancer. The procedure involves taking a cheek swab, which is then analysed using non-damaging infrared light technology.

The RADICAL REACT study To introduce this technology into a healthcare setting the sponsor needs to validate its effectiveness through rigorous testing.

The RADICAL REACT trial plans to involve around 450 participants highly suspected to have lung cancer. Each participant will provide a cheek swab and basic medical history information during a single clinic visit. The data collected will be analysed with AIR-DS to identify whether individuals with lung cancer can be identified accurately.

Why it matters AIR-DS could significantly advance lung cancer detection, focusing on early, accurate diagnosis through a non-invasive cheek swab. Beyond improving patient outcomes by enabling timely intervention, it also introduces a cost-effective approach to early lung cancer detection. AIR-DS aims to alleviate the financial burden on healthcare systems and patients by reducing the need for more expensive and/or invasive diagnostic procedures.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, study participants must meet all the following criteria:

* Can understand and provide signed consent.
* Are aged 18 years or older.
* Can provide a cheek swab sample.
* Are symptomatic of, and/or are being investigated for, lung cancer.
* Have not commenced treatment for lung cancer.

Exclusion Criteria:

Study participants who meet any of the following criteria will be excluded from participation in this study:

* Are pregnant.
* Have been diagnosed with another known malignancy within five years (excluding localised squamous cell carcinoma of the skin, cervical intraepithelial neoplasia, grade III and low-grade prostate cancer (Gleason score <5 with no metastases)).
* Have a concurrent disease, medical condition, or extenuating circumstances that, in the opinion of the investigator, might compromise study completion or data collection, including:

  1. Localised oral disease, including but not limited to periodontitis, bleeding gums, dysplastic mouth disease.
  2. Taking anti-coagulants.
  3. Alpha 1 anti-trypsin deficiency.
  4. Active infections such as tuberculosis.
  5. Conditions that in the opinion of the investigator are not controlled e.g. hypertension, asthma, chronic kidney disease, bowel disease, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 450 participants will be recruited into the study from at risk or symptomatic patients being evaluated for lung cancer. The study aims to recruit approximately 196 participants with lung cancer. Recruitment will be continually monitored and may be stopped earlier than planned if the investigators have recruited 196 participants with lung cancer and with a sufficient proportion of early-stage lung cancer.
  Participants who withdraw or are deemed a screen failure will be replaced and will not count towards the overall recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Day 1
  Evaluate the sensitivity of AIR-DS pre-specified algorithm in identifying lung cancer when compared to a clinical diagnosis in a high-incidence lung cancer population.

SECONDARY OUTCOMES:
Specificity, PPV, NPV | Day 1
  Evaluate the specificity, positive and negative predictive values of AIR-DS pre-specified algorithm in identifying lung cancer compared to a clinical diagnosis of lung cancer, in a high-incidence lung cancer population.
Predictive performance of refined predictive algorithm | 12 months after the last participant is recruited
  Predictive performance (e.g. accuracy, sensitivity, specificity, NPV, PPV, AUC) classifying lung cancer as compared with a clinical diagnosis, in a high-risk lung cancer population using the updated algorithm following refinement of the predictive algorithm and cutting points of AIR-DS
Performance of predictive algorithm across lung cancer type and stage | Day 1
  Predictive performance (e.g. accuracy, sensitivity, specificity, NPV, PPV) of AIR-DS pre-specified algorithm compared to a clinical diagnosis of lung cancer in participants with: no lung cancer vs. NSCLC; no lung cancer vs. SCLC; no lung cancer vs. stage 1 lung cancer; and no lung cancer vs. stage 2 lung cancer.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Northumbria Healthcare NHS Foundation Trust, North Shields
  - Queen Alexandra Hospital, Portsmouth

IPD SHARING:
Plan to Share IPD: Undecided
To be decided